CLINICAL TRIAL: NCT01492023
Title: The Effects of Attention Retraining on Cognitive Performance, QoL and Perceived Cognitive Impairment in MS - a Single Blind, Randomized, Controlled Study
Brief Title: The Effects of Attention Retraining in MS
Acronym: MSattention
Status: Completed | Type: Observational
Sponsor: Finnish MS Society (Other)
Collaborators: Social Insurance Institution, Finland (Other); Tampere University Hospital (Other); Seinajoki Central Hospital (Other)
Responsible Party: Principal Investigator, Paivi Hamalainen, neuropsychologist, adjunct professor, Finnish MS Society
Other Study IDs: MS1209
Record Dates: First submitted 2011-12-04; First posted 2011-12-14 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Sclerosis
Keywords: neuropsychological; rehabilitation; multiple sclerosis; RCT study
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — A randomised, controlled, single-blind study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: control group: no intervention
- neuropsychological rehabilitation: intervention group: neuropsychological rehabilitation (13 times 60 minutes, once per week, during 13 weeks) control group: no intervention
  Interventions: Behavioral: neuropsychological rehabilitation

INTERVENTIONS:
Behavioral: neuropsychological rehabilitation — attention retraining and teaching compensatory strategies as well as offering psychological support to better cope with cognitive impairments (13 times 60 minutes, once per week during 13 weeks)
  Groups: neuropsychological rehabilitation

SUMMARY:
The purpose of this study is to determine whether neuropsychological rehabilitation focused on attention retraining and teaching compensatory strategies has positive effects on cognitive performance, quality of life (QoL)and perceived cognitive deficits in patients with MS. The hypothesis is that the neuropsychological intervention shows positive effects on cognitive performance, QoL and perceived cognitive deficits.

DETAILED DESCRIPTION:
Background: Cognitive impairments are a typical manifestation of multiple sclerosis (MS). According to previous studies, neuropsychological rehabilitation may improve cognitive performance in MS. However, the quality of previous studies is low and, accordingly, the evidence on the effects of neuropsychological rehabilitation is low to modest.

Objective: To study whether neuropsychological rehabilitation improves cognitive performance, QoL and perceived cognitive deficits in patients with MS.

Methods: Altogether 100 patients with MS are randomised either to intervention or to control group in three different study sites. All the study subjects are assessed with neuropsychological tests as well as self-rating questionnaires evaluating mood, QoL, cognitive deficits, fatigue and impact of the disease at baseline, after three months (immediately after intervention) and after six months. Patients in the intervention group are offered with neuropsychological rehabilitation conducted once a week during thirteen weeks. Patients in the control group do not receive any intervention.

Results: The effects of intervention on cognitive performance, QoL and perceived cognitive impairments are evaluated using appropriate statistical procedures and comparing the differences between the intervention and the control group.

The present status: The baseline assessments have been performed and the intervention will be conducted between September and December, 2011.

ELIGIBILITY:
Inclusion Criteria:

* clinically definite MS
* EDSS < 6
* age 18-58 years
* subjective cognitive problems and objective decline in attention

Exclusion Criteria:

* other neurological disease than MS
* psychiatric diagnosis
* severe depression
* secondary progressive or primary progressive course of MS
* EDSS>=6
* alcohol or drug abuse
* relapse during the preceding month of study entry
* neuropsychological rehabilitation during the study
* no subjective cognitive cognitive problems and /or no decline in attention
* overall cognitive impairment (performance in all tests of BRBNT under -1.5 SD compared to norms of healthy controls)

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with MS are collected from community by informing about the study via information letters send to the members of local MS Associations
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Objective cognitive performance | six months
  effects of rehabilitation on objective cognitive performance: SDMT
Subjective cognitive performance | six months
  The effects of rehabilitation on subjective cognitive performance: perceived cognitive deficits (Perceived Deficits Questionnaire, PDQ)
Goal achievement | six months
  Goal achievement: Goal Attainment Scaling (GAS)

SECONDARY OUTCOMES:
Quality of life | six months
  The effects of rehabilitation on QoL: WHOQOL-Bref
Objective cognitive performance | six months
  The effects of rehabilitation on cognitive performances: test of Brief Repeatable Battery of Neuropsychological Tests (BRBNT), Trail Making Test, Stroop test
Mood | six months
  The effects of rehabilitation on mood: Beck Depression Inventory II (BDI II)
Fatigue | six months
  The effects of rehabilitation on self-perceived feeling of fatigue: Fatigue Scale for Motor and Cognitive Fatigue (FSMC)
Subjective cognitive performance | six months
  The effects of rehabilitation on subjective cognitive performance evaluated by the patient him/herself or the significant other: Multiple Sclerosis Neuropsychological Questionnaire (MSNQ-P, MSNQ-I)
The impact of the disease | six months
  The effects of rehabilitation on the impact of the disease: Multiple Sclerosis Impact Scale (MSIS-29)

CONTACTS AND LOCATIONS:
Overall Officials: Päivi I Hämäläinen, adjunct prof, Study Director — Finnish MS Society / Masku Neurological Rehabilitation Centre; Keijo Koivisto, Prof, Study Chair — Seinajoki Central Hospital; Eija M Rosti-Otajärvi, PhD, Principal Investigator — Tampere University Hospital; Anu Mäntynen, MA, Principal Investigator — Seinajoki Central Hospital
Locations (3):
- Finland (3):
  - Masku Neurological Rehabilitation Centre, Masku
  - Seinajoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere